CLINICAL TRIAL: NCT01261988
Title: A Single Center, Feasibility Study Using Healthy Volunteers to Assess the Safety and Adhesive Performance of the VIPER System When Compared to the Esteem™ Cut to Fit One Piece Closed End Pouch
Brief Title: Assess the Safety and Adhesive Performance of the VIPER System When Compared to Esteem™
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Qing Li, Assoc Dir Clinical Research, Convatec Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-0512-10-A723
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2010-12-20 (Estimated); Status verified 2010-12

CONDITIONS: Ostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: VIPER — Comparison of ostomy systems
Device: Esteem™ Cut to Fit One Piece Closed End Pouch — Comparison of ostomy systems

SUMMARY:
The primary objective of the study is to assess the safety and adhesive performance of the VIPER System when compared to the Esteem™ Cut to Fit One Piece Closed End Pouch when used by healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 70 years of age (inclusive) at the time of randomization
* Willing and able to provide written informed consent and HIPAA Waiver
* An appropriate candidate for participation with unbroken non-irritated abdominal skin
* Willing to adhere to the study procedures and to attend the scheduled study visits according to the requirements of the study protocol
* Willing to adhere to the scheduled study visits
* Good manual dexterity and be able to take care of their abdominal area independently
* Be willing and able to record the required study data in a specified format

Exclusion Criteria:

* A history of a known sensitivity or allergy to System 3+ adhesive (modified Stomahesive® technology), Stomahesive®, Durahesive®, Polyethylene Film, or polyester fiber,or to any adhesive components in general as listed in the Investigators Brochure.
* Subjects who have any other medical condition which, according to the investigator justifies exclusion from the study
* Subjects with any chronic allergies requiring the use of prescription medication
* History of skin disease affecting abdominal area
* Currently uses topical ointments in the area of the abdomen or is unwilling/unable to terminate over the counter use of topical ointments in the area of the abdomen
* Active case of eczema, dermatitis, psoriasis
* Pregnant or lactating females.
* Subject currently enrolled in another investigational study
* Possesses extensive knowledge about either product (ie employees that re members or extended members of the Core Team work in ostomy research and development, or ostomy division sales and marketing )

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety: Related Events | 17 hours
  All adverse events (AE's) related to the use of the device
Efficacy: Device Fall-Offs | 17 hours
  The number and percentage of subjects with study device fall-off during the study
Efficacy: Device Fall-Offs | 17 hours
  The total number of study device fall-offs during the course of the study
Safety: Skin Reactions | 17 hours

SECONDARY OUTCOMES:
Adhesive | 1 hour
  Initial tack of the adhesive (during first hour of wear)
Ease of Removal | 17 hours
  Ease of removal of the adhesive wafer from the skin
Security | 17 hours
  Perceived security of the study pouch during wear

CONTACTS AND LOCATIONS:
Overall Officials: Qing Li, PhD, Study Director — ConvaTec Inc.
Locations (1):
- Susan Bell, RN, MSN, CWOCN, Jobstown, New Jersey, United States